CLINICAL TRIAL: NCT04016961
Title: Huma-Animal Interaction to Promote Recovery Following Pediatric Brain Injury
Brief Title: Human-Animal Interaction to Promote Recovery Following Pediatric Brain Injury
Acronym: AAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CIN001-AAT; 1R21HD095132-01 (NIH)
Record Dates: First submitted 2019-05-03; First posted 2019-07-12 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Brain Injuries; Acquired Brain Injury; Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animal Assisted Therapy - Dog Session (Experimental): Therapy dog added to PT and OT session
  Interventions: Other: AAT - Dog
- Treatment as usual - No Dog session (Active Comparator): No dog added to PT and OT session - PT and OT session as usual standard of care
  Interventions: Other: TAU - No Dog

INTERVENTIONS:
Other: AAT - Dog — therapy dog added to inpatient PT and OT session
  Arms: Animal Assisted Therapy - Dog Session
Other: TAU - No Dog — PT and OT as usual without the addition of therapy dog
  Arms: Treatment as usual - No Dog session

SUMMARY:
This study evaluates the addition of therapy dogs in inpatient physical and occupational therapy. Data will be collected across 10 PT and 10 OT sessions, half of which will incorporate a therapy dog.

DETAILED DESCRIPTION:
Children with acquired brain injuries (ABI) treated on an inpatient rehabilitation unit are at significant risk for long term functional impairment, highlighting the importance of maximizing the effectiveness and utilization of inpatient rehabilitation therapies. The proposed study seeks to explore the value of animal-assisted therapy (AAT) during inpatient rehabilitation following pediatric ABI. Investigators will employ a within subjects cross-over trial; all participants will have a volunteer dog involved in 50% of their physical therapy (PT) and occupational therapy (OT) sessions over a 2-week study period. AAT will consist of integration of a dog from the hospital volunteer dog program in PT and OT sessions, while the non-AAT condition will be treatment as usual (TAU) as identified by the patients' treatment team. Information regarding patient engagement/participation in therapy, affect, and physiological variables will be collected during each session. Session notes will also be coded for additional qualitative information. Qualitative feedback from patients and families, therapists, medical teams, and dog handlers will also be collected throughout the project to examine feasibility and satisfaction with the intervention as well as potential barriers and areas for improvement. Investigators will 1) examine the effect of AAT on level of patient participation and patient affect during PT and OT sessions, 2) Explore the effect of AAT on functional outcomes using a historic cohort comparison group, and 3) explore the physiological response of patients, and examine a number of variables (injury type/severity, child sex and anthropomorphism, therapist factors, and dog handler factors) to begin to determine which patients are most likely to benefit from AAT during inpatient rehabilitation for ABI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Participants must be on the inpatient rehabilitation unit for treatment of an acquired brain injury (TBI, brain tumor, infection, stroke, etc)
* Consent: The family must provide informed consent by parents or legal guardians
* Assent: The adolescent must provide a signature indicating assent to participate in the study.
* Age at time of screening: 6 years old and older with no upper limit
* Responsiveness: Rancho score greater than 2 (or equivalent) at the time of enrollment (as noted in medical chart)

Exclusion Criteria:

* Animals: Participant has a significant allergy to dogs or have a significant fear of dogs.
* Disease: Participant has a communicable disease that may pose a risk to dog or dog handler or a compromised immune system where interacting with dog and/or handler would be of significant risk to patient.
* Responsiveness: Rancho score of 2 (or equivalent) or less
* Cognitive issues: Participants with pre-injury/pre-diagnosis of developmental delay, autism, and/or patients who are non-verbal will be excluded.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Patient Participation - AAT | Throughout study completion, an average of 2 weeks
  Patient participation during AAT sessions will be assessed using the Pittsburgh Rehabilitation Participation Scale (PRPS)The PRPS is a 6-item Likert-type, clinician-rated measure that quantifies observed patient participation in their therapy session. Therapists report their observations regarding patient's completion of exercises, effort applied to exercises, and level of support needed to complete activities. Scores range from 1 (None) to 6 (excellent). Therapists will complete this measure at the end of each AAT session. Ratings across the 5 (on average) AAT sessions will be used to create an patient participation - AAT score.
Patient Participation - TAU | Throughout study completion, an average of 2 weeks
  Patient participation during TAU sessions will be assessed using the Pittsburgh Rehabilitation Participation Scale (PRPS)The PRPS is a 6-item Likert-type, clinician-rated measure that quantifies observed patient participation in their therapy session. Therapists report their observations regarding patient's completion of exercises, effort applied to exercises, and level of support needed to complete activities. Scores range from 1 (None) to 6 (excellent). Therapists will complete this measure at the end of each TAU session. Scores across the 5 (on average) TAU sessions will be used to create a single patient participation - TAU score.
Objective session participation - AAT | Throughout study completion, an average of 2 weeks
  Objective session participation will be assessed via videotaped sessions for at least 2 AAT sessions. Coders will provide an objective measure of participation by rating patient in session participation using the Pittsburgh Rehabilitation Participation Scale (PRPS). Coders will score participation using the PRPS and rate the participants level of participation from 1 (None) to 6 (Excellent). These coder ratings will be used to create an overall objective session participation AAT score.
Objective session participation - TAU | Throughout study completion, an average of 2 weeks
  Objective session participation will be assessed via videotaped sessions for at least 2 TAU sessions. Coders will provide an objective measure of participation by rating patient in session participation using the Pittsburgh Rehabilitation Participation Scale (PRPS). Coders will score participation using the PRPS and rate the participants level of participation from 1 (None) to 6 (Excellent). These coder ratings will be used to create an overall objective session participation TAU score.
Patient Affect - AAT | Throughout study completion, an average of 2 weeks
  Patient affect will be assessed via the Symptom Inventory Scale - Short.This measure is a 4-item measure, where the patient reports the degree (from 0-10) they are experiencing each feeling/condition presented (Happy, fatigue, distraction, irritability). The patient will be asked to complete this measure at the beginning and end of each AAT session. These ratings will be used to create happy, fatigue, distracted, and irritable - AAT scores. Greater scores are reflective of greater levels of that emotion.
Patient Affect - TAU | Throughout study completion, an average of 2 weeks
  Patient affect will be assessed via the Symptom Inventory Scale - Short.This measure is a 4-item measure, where the patient reports the degree (from 0-10) they are experiencing each feeling/condition presented (Happy, fatigue, distraction, irritability). The patient will be asked to complete this measure at the beginning and end of each TAU session. These ratings will be used to create happy, fatigue, distracted, and irritable - TAU scores. Greater scores are indicative of greater levels of that emotion.
Objective mood assessment - AAT | Throughout study completion, an average of 2 weeks
  Objective mood assessment will be completed for at least 2 AAT sessions via coding of video taped sessions. Coders naïve to hypotheses will assess the percentage of time the patient displays positive and negative affect. Greater scores. Greater scores are indicative of greater levels of positive and negative affect. Scores across all coded AAT sessions will be used to create a positive affect-AAT score and negative affect-AAT score.
Objective mood assessment - TAU | Throughout study completion, an average of 2 weeks
  Objective mood assessment will be completed for at least 2 TAU sessions via coding of video taped sessions. Coders naïve to hypotheses will assess the percentage of time the patient displays positive and negative affect. Greater scores. Greater scores are indicative of greater levels of positive and negative affect. Scores across all coded TAU sessions will be used to create a positive affect-TAU score and negative affect-TAU score.

SECONDARY OUTCOMES:
Heart rate- AAT | Throughout study completion, an average of 2 weeks
  Heart rate will be collected using an Empatica E4 wristband during each of the AAT sessions. The patient will wear the wrist band during all sessions, and data collected during AAT sessions will be summarized as heart rate - AAT,
Temperature - AAT | Throughout study completion, an average of 2 weeks
  Temperature will be collected using an Empatica E4 wristband during each of the AAT sessions. The patient will wear the wrist band during all sessions, and data collected during AAT sessions will be summarized as temperature-AAT.
Galvanic Skin Response - AAT | Throughout study completion, an average of 2 weeks
  Galvanic skin response (GSR) will be collected using an Empatica E4 wristband during each of the AAT sessions. The patient will wear the wrist band during all sessions, and data collected during AAT sessions will be summarized as GSR-AAT.
Heart Rate - Tau | Throughout study completion, an average of 2 weeks
  Heart rate will be collected using an Empatica E4 wristband during each of the TAU sessions. The patient will wear the wrist band during all sessions, and data collected during TAU sessions will be summarized as heart rate - TAU.
Temperature - Tau | Throughout study completion, an average of 2 weeks
  Temperature, and galvanic skin response will be collected using an Empatica E4 wristband during each of the TAU sessions. The patient will wear the wrist band during all sessions, and data collected during TAU sessions will be summarized as temperature-TAU.
Galvanic skin response - Tau | Throughout study completion, an average of 2 weeks
  Galvanic skin response (GSR) will be collected using an Empatica E4 wristband during each of the TAU sessions. The patient will wear the wrist band during all sessions, and data collected during TAU sessions will be summarized as GSR-TAU.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Narad, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No